CLINICAL TRIAL: NCT04095273
Title: A Multicenter, Non-randomized, Open-label Phase 1b Study to Determine the Maximum Tolerated and Recommended Phase 2 Dose of the ATR Inhibitor Elimusertib in Combination With Pembrolizumab and to Characterize Its Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity in Participants With Advanced Solid Tumors
Brief Title: Study to Test How Well Patients With Advanced Solid Tumors Respond to Treatment With the Elimusertib in Combination With Pembrolizumab, to Find the Optimal Dose for Patients, How the Drug is Tolerated and the Way the Body Absorbs, Distributes and Discharges the Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19741; KEYNOTE-919 (Other: Merck); MK-3475-919 (Other: Merck); 2018-003420-36 (EudraCT Number)
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumors
Keywords: DDR (Deoxyribonucleic acid damage repair),; ATR (ataxia-telangiectasia and Rad3 related protein)inhibitor,
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Ataxia Telangiectasia | interventions — BAY 1895344; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Dose escalation of Elimusertib (Experimental): 2 dose levels of Elimusertib are planned
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 1a of Elimusertib (Experimental): Participants with advanced hormone-receptor-positive, Human epidermal growth factor receptor 2 negative breast cancer (HER2-negative BC), known to be positive for Ataxia-telangiectasia mutated (ATM) loss and/or ATM deleterious alterations who have not received prior treatment with immunotherapy. Participants with known microsatellite instability-high (MSI-H) cannot be included
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 1b of Elimusertib (Experimental): Participants with advanced hormone-receptor-positive, HER2-negative BC, known to be DDR deficiency biomarker-positive (except ATM loss/mutation) who have not received prior treatment with immunotherapy. Participants with known MSI-H cannot be included.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 2a of Elimusertib (Experimental): Participants with advanced Colorectal cancer (CRC) known to be positive for ATM loss and/or ATM deleterious alterations who have not received prior treatment with immunotherapy. Participants with known MSI-H cannot be included.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 2b of Elimusertib (Experimental): Participants with advanced CRC, known to be DDR deficiency biomarker -positive (except ATM loss/mutation) who have not received prior treatment with immunotherapy. Participants with known MSI-H cannot be included.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 3 of Elimusertib (Experimental): Participants with advanced Gastric/gastroesophageal junction cancer (GC/GEJ) known to be DDR deficiency biomarker-positive (incl. ATM mutation) and/or positive for ATM loss. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 3a of Elimusertib (Experimental): Participants with advanced GC/GEJ cancer and without DDR deficiency alterations as described above. Variants of unknown significance (VUS) of the DDR gene alterations are eligible. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 4 of Elimusertib (Experimental): Participants with advanced Non-small cell lung cancer (NSCLC) known to be DDR deficiency biomarker-positive (incl. ATM mutation) and/or positive for ATM loss. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 4a of Elimusertib (Experimental): Participants with advanced NSCLC and without DDR deficiency alterations as described above. VUS of the DDR gene alterations are eligible. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 5 of Elimusertib (Experimental): Participants with advanced pancreatic cancer, known to be DDR deficiency biomarker-positive (incl. ATM mutation) and/or positive for ATM loss who have not received prior treatment with immunotherapy. Participants with known MSI-H cannot be included.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 5a of Elimusertib (Experimental): Participants with advanced pancreatic cancer and without DDR deficiency alterations as described above, who have not received prior treatment with immunotherapy. VUS of the DDR gene alterations are eligible. Participants with known MSI-H cannot be included.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 6 of Elimusertib (Experimental): Participants with advanced Metastatic castration-resistant prostate cancer (mCRPC), known to be DDR deficiency biomarker positive (incl. ATM mutation) and/or positive for ATM loss who have not received prior treatment with immunotherapy. Participants with known MSI-H cannot be included.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)
- Dose expansion cohort 6a of Elimusertib (Experimental): Participants with advanced mCRPC and without DDR deficiency alterations as described above, who have not received prior treatment with immunotherapy. VUS of the DDR gene alterations are eligible. Participants with known MSI-H cannot be included.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Pembrolizumab (Keytruda®)

INTERVENTIONS:
Drug: Elimusertib (BAY1895344) — Study drugs will be administered as scheduled
Drug: Pembrolizumab (Keytruda®) — Study drugs will be administered as scheduled

SUMMARY:
The purpose of the study is to test how well patients with advanced solid tumors respond to treatment with elimusertib (BAY1895344) in combination with pembrolizumab. In addition researchers want to find for patients the optimal dose of elimusertib in combination with pembrolizumab, how the drug is tolerated and the way the body absorbs, distributes and discharges the drug. The study medication, elimusertib, works by blocking a substance (ATR Kinase) which is produced by the body and is important for the growth of tumor cells. Pembrolizumab is an immunologic checkpoint blocker that promotes an immune response against the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age inclusive, at the time of signing the informed consent.
* Presence of the putative biomarkers of DDR deficiency in tumor and/or other tissues (dose escalation only).
* Participants must have histologically confirmed solid tumors .
* Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 to 1.
* Adequate bone marrow function as assessed by laboratory tests to be conducted within 7 days before the first dose of study intervention.
* Participants must have adequate kidney function, as assessed by the estimated glomerular filtration rate (eGFR) > 40 mL/min per 1.73 m*2 within 7 days before the first dose of study intervention.
* Participants must have adequate liver function as assessed by laboratory tests to be conducted within 7 days before the first dose of study intervention.
* Participants must have adequate coagulation, as assessed by laboratory tests as applicable, (to be conducted within 7 days before the first dose of study intervention) or be on stable anti-coagulation treatment.
* Adequate cardiac function per institutional normal measured by echocardiography (recommended) or multigated acquisition (MUGA) scan/cardiac MRI per institutional guidelines.
* Participants must have measurable disease (at least one measurable lesion) as per RECIST 1.1, or evaluable disease according to the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) classification as applicable. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions

Exclusion Criteria:

* Ongoing infections of Common terminology criteria for adverse events (CTCAE) grade ≥2 not responding to therapy or active clinically serious infections.
* Participants with

  * Known human immunodeficiency virus (HIV)
  * Active Hepatitis B infection (positive for Hepatitis B surface antigen (HBsAg)/ Hepatitis B virus (HBV) DNA).
  * Active Hepatitis C infection (positive anti-HCV Antibody and quantitative HCV RNA results greater than the lower limits of detection of the assay).
* Active autoimmune disease (active defined as having autoimmune disease related symptoms and detectable autoantibodies) that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Diagnosis of immunodeficiency or participant is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention. The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor.
* Pleural effusion or ascites that causes respiratory compromise (CTCAE Grade ≥ 2 dyspnea).
* History of cardiac disease: congestive heart failure New York Heart Association (NYHA) class >II, unstable angina (angina symptoms at rest), new-onset angina (within the past 6 months before study entry), myocardial infarction within the past 6 months before study entry, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers, calcium channel blockers, and digoxin are permitted)
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's opinion)
* Moderate or severe hepatic impairment, i.e., Child-Pugh class B or C.
* History of organ allograft transplantation
* Evidence or history of bleeding disorder, i.e., any hemorrhage / bleeding event of CTCAE Grade > 2 within 4 weeks before the first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) including Treatment Emergent Serious Adverse Events (TESAEs) | Up to 30 days after last study intervention administration
Severity of Treatment Emergent Adverse Events (TEAEs) including Treatment Emergent Serious Adverse Events (TESAEs) | Up to 30 days after last study intervention administration
Frequency of Dose limiting toxicities (DLTs) at each dose level during dose escalation of BAY1895344 | Cycle 1 (21 days)
Recommended phase II dose (RP2D) of BAY1895344 | Up to 24 months
  The RP2D will be determined in dose expansion part based on multiple parameters (i.e., safety, tolerability, PK, pharmacodynamics, efficacy) and will be a dose equal to or lower than the MTD (Maximum Tolerated Dose).

SECONDARY OUTCOMES:
Cmax of Elimusertib | Cycle 1 (21 days), Day 8 (dosing schedule 1) or Cycle 1 (21 days), Day 1 (dosing schedule 2)
AUC(0-12) of Elimusertib | Cycle 1 (21 days), Day 8 (dosing schedule 1) or Cycle 1 (21 days), Day 1 (dosing schedule 2)
  If the main parameters AUC(0-12) cannot be calculated reliably, it might become necessary to appoint the additional parameters AUC(0-tlast) as secondary variables.
Cmax,md of Elimusertib | Cycle 1 (21 days), Day 17 (dosing schedule 1) or Cycle 1 (21 days), Day 10 (dosing schedule 2)
AUC(0-12)md of Elimusertib | Cycle 1 (21 days), Day 17 (dosing schedule 1) or Cycle 1 (21 days), Day 10 (dosing schedule 2)
  If the main parameters AUC(0-12)md cannot be calculated reliably, it might become necessary to appoint the additional parameters AUC(0-tlast)md as secondary variables.
Incidence of Complete response (CR) | Up to 24 months
  Per RECIST 1.1 and for participants with mCRPC consistent with recommendations of the Prostate Cancer Working Group (PCWG3)
Incidence of partial response (PR) | Up to 24 months
  Per RECIST 1.1 and for participants with mCRPC consistent with recommendations of the Prostate Cancer Working Group (PCWG3)
Incidence of stable disease (SD) | Up to 24 months
  Per RECIST 1.1 and for participants with mCRPC consistent with recommendations of the Prostate Cancer Working Group (PCWG3)
Incidence of progressive disease (PD) | Up to 24 months
  Per RECIST 1.1 and for participants with mCRPC consistent with recommendations of the Prostate Cancer Working Group (PCWG3)
Objective Response Rate (ORR) | Up to 24 months
Disease control rate (DCR) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (8):
  - Stanford University, Palo Alto, California
  - Yale Cancer Center, New Haven, Connecticut
  - Johns Hopkins Hospital/Health System, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (2):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Eberhard-Karls-Universität Tübingen, Tübingen, Baden-Wurttemberg
- Spain (2):
  - Fundacion Jimenez Diaz (Clinica de la Concepcion), Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
- Switzerland (2):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Ospedale Regionale di Bellinzona e Valli, Bellinzona, Canton Ticino
- United Kingdom (2):
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - Freeman Hospital, Newcastle, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/19741